CLINICAL TRIAL: NCT03456765
Title: Fetal Kidney in Estimation of GA and Maturity
Brief Title: Fetal Kidney in Estimation of GA in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other); National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: fetal kidney
Record Dates: First submitted 2018-03-05; First posted 2018-03-07 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Gestational Age and Maturity
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — US will be made to assess kidneys

SUMMARY:
A true estimation of gestational age (GA) plays animportant role in quality of maternity care such asassessment of fetal growth and to schedule the labordate. Any inaccurate estimation may lead to peri-natalmorbidity and mortality due to iatrogenic pre- or post-maturity .

DETAILED DESCRIPTION:
Several longitudinal studies have been performed in the western countries concerning sonographic measurement of fetal kidney length. Initially these were done for diagnosis of renal malformation in utero & later on they were to find out the correlation between the fetal kidney length and the gestational age

ELIGIBILITY:
Inclusion Criteria:

1. Single fetus.
2. pregnant ladies. with no medical disorders
3. Fetal kidneys are normally seen

Exclusion Criteria:

* Medical disorders with pregnancy
* Renal anomalies
* Renal agesnesis

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females
Study Population: pregnant ladies with no medical disorders with pregnancy between 16 weeks and 40 weeks in a single living fetus
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-04-20 (Estimated)

PRIMARY OUTCOMES:
The number of participants who will have accurate GA calculated by Kidney parameters | within 2 months
  describes the efficiency of kidney parameters to estimate GA

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt